CLINICAL TRIAL: NCT04028661
Title: Evaluation of 3D Printed Modified Twin Block Appliance for Correction of Skeletal Class II Malocclusion in Growing Subjects: A Randomized Controlled Trial
Brief Title: Evaluation of 3D Printed Modified Twin Block for Correction of Skeletal Class II Malocclusion in Growing Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, : Donia Ayman Ahmed Ezzeldin ElSayed, Master degree student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1993
Record Dates: First submitted 2019-07-15; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Class II Malocclusion, Division 1
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Intervention Model Description: The design of this randomized controlled trial is a parallel group, two arm, superiority trial with 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, the operator and patients can't be blinded. Blinding of the outcome assessors can be done by sealing the name of the patient and the of the pre and post treatment radiographs used for analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): use of 3D printed Modified Twin Block Appliance.
  Interventions: Device: 3D printed Modified Twin Block Appliance
- Untreated control group (No Intervention): No treatment phase of 8 months.

INTERVENTIONS:
Device: 3D printed Modified Twin Block Appliance — It is a functional appliance for mandibular advancement designed digitally on virtual models.
  Arms: Intervention group

SUMMARY:
The study is to evaluate the effect of 3D printed modified Twin Block Appliance on skeletal Class II profile correction.

The null hypothesis of this research is that use of 3D Printed Twin Block is not able to induce skeletal rather than dental effects for correction of the skeletal Class II malocclusion in comparison with untreated growing Class II control subjects.

DETAILED DESCRIPTION:
I- For the treatment group:

A- Medical History Questionnaire will be filled by the patient to exclude the presence of any systemic condition.

B- Clinical Examination:

Proper examination of the oral structures including;

* Teeth will be examined for caries, fracture or missing teeth
* Gingival tissues will be examined for gingivitis, periodontitis, attachment loss, gingival recession, oral lesions and the nature of the gingival biotype.
* Thorough intraoral examination is needed to evaluate the need for referral for consultation or intervention before the initiation of treatment.

C- Diagnosis:

* The patient is checked to fulfil the inclusion criteria.
* A clinical visualized treatment outcome (VTO) will be done by asking the patient to bite in an advanced position and check the outcome of this advancement on the patient"s profile. Patients with positive results (better profiles were achieved upon advancement) are included in the study.
* Full set of records (including standardized Lateral Cephalograms) will be taken for every 8 patient as part of the routine procedure for treatment of patients in the outpatient clinic of the Orthodontic Department, Cairo University.

D- Clinical Procedures:

After taking upper and lower impressions, the impressions are then poured into hard stone that are then digitally scanned using 3D laboratory scanner (3Shape R500 Lab Scanner).

Designing the appliance is done on upper and lower virtual models (using 3Shape Appliance Designer). The appliance covers the upper and lower dental arches with lingual horizontal rectangular attachments to increase the retention.

Buccal triangular ramps for mandibular advancement are designed. They are positioned buccal to the upper and lower posterior segments with a lock to ensure the desired mandibular advancement.

3D printing of the appliance is then done using 3D printer (Dent2-Mogassam) with biocompatible resin material (NextDent Resin OrthoRigid).

Post curing using ultraviolet light for 30min using postcuring unit (Postcuring- Mogassam).

The appliance is then delivered to the patient and instructions are given. Follow up every 4 weeks for 8 months or edge to edge occlusion (the sooner) and then full records taken including Lateral Cephalogram.

II- For the Control group

* The subjects should be fulfilling the previously mentioned inclusion criteria and should sign the informed consent of agreement to be recruited in the study.
* According to the randomization sheet, the patients allocated to the control group will be immediately referred for the uptake of a Lateral Cephalogram which will be considered (T1) without any treatment procedures.
* A "no treatment" phase of 8 months will be carried out through which the patients will be followed up to monitor any factor that might have occurred to exclude the patient from the study.
* Another Lateral Cephalogram will be taken after 8 months (T2).
* T2 images are to be considered the initial diagnostic images for the patient. The patients will be then assessed and treatment will be provided for each patient as required.

ELIGIBILITY:
Inclusion Criteria:

* Females 10-13 years of age.
* Skeletal Angle Class II division 1 malocclusion with a deficient mandible. (SNB ≤ 76°)
* Horizontal or neutral growth pattern. (MMP ≤ 30°)
* Increased overjet (min 5 mm) with Class II canine relationship. (minimum of half unit)
* Cervical Vertebral Maturation (CVM) stage 3.

Exclusion Criteria:

* Systemic Disease.
* Any signs or symptoms or previous history of temporomandibular disorders (TMD) as clicking, crepitus, pain, limitation or deviation.
* Extracted or missing upper permanent tooth/teeth (except for third molars).
* Facial Asymmetry.
* Para-functional habits.
* Severe proclination or crowding that requires extractions in the lower arch.

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Skeletal Class II profile correction | 8months
  A-Effective mandibular length in mm B- SNB in degrees using lateral cephalogram

SECONDARY OUTCOMES:
Inclination of anterior teeth | 8 months
  A- L1/MP in degrees using lateral cephalogram B- L1-FP in mm
Soft tissue convexity correction | 8 months
  Angle of convexity (N"-Sn/ N"-Pog") in degrees using lateral cephalogram
Patient acceptance | 8 months
  Five point Likert scale is used to allow the individual to express how much they agree or disagree with a particular statement.
  Points of Scale 5 (very satisfied) (the best) 4 (satisfied) 3 (Neutral) 2 (Dissatisfied)
  1 (Very Dissatisfied) (the worst)

CONTACTS AND LOCATIONS:
Overall Officials: Donia Ezzeldin, Master, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No